CLINICAL TRIAL: NCT02546726
Title: Heat & Aerobic Training (HEAT) for Pre-Hypertensive Middle-Aged Adults
Brief Title: Heat & Aerobic Training (HEAT) Study
Acronym: HEAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Urbana-Champaign (Other)
Responsible Party: Principal Investigator, Sean Mullen, Associate Professor of Kinesiology & Community Health, University of Illinois at Urbana-Champaign
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RB15229; 15935 (Other: UIUC Institutional Review Board)
Record Dates: First submitted 2015-08-18; First posted 2015-09-11 (Estimated); Last update posted 2019-04-17 (Actual); Status verified 2019-04

CONDITIONS: Pre-hypertension
Keywords: heat therapy; steam-room; aerobic exercise; hypertension; multiple behavior change; lifestyle modification
MeSH Terms: conditions — Prehypertension; Hyperthermia; Hypertension | interventions — Hot Temperature; Steam

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Heat & Aerobic Training (HEAT) Condition (Experimental): Participants will receive supervised, moderate intensity (50-75% maximum heart rate) aerobic exercise sessions, 3 times per week for 50 minutes in duration. After the exercise portion of each session, participants assigned to the HEAT condition will be asked to sit quietly on the bench in the steam-room within their same-sex locker room for no more than 20 minutes. They will start at 11 minutes to get acclimated to the mild heat stress, and gradually work up to 20 minutes. A trained research staff member will be stationed outside the room.
  Interventions: Behavioral: Heat & Aerobic Training (HEAT)
- Exercise Only (Active Comparator): Participants will receive supervised, moderate intensity (50-75% maximum heart rate) aerobic exercise sessions, 3 times per week for 50 minutes in duration. After the exercise portion of each session, participants assigned to the Exercise Only condition will be asked to sit quietly on the bench in the lobby of the fitness facility, initially for 11 minutes and then gradually working up to 20 minutes.
  Interventions: Behavioral: Exercise Only

INTERVENTIONS:
Behavioral: Heat & Aerobic Training (HEAT) — Participants receive 42 supervised 50-minute, moderately intensive (50-75% max HR) aerobic exercise sessions (3 times per week), followed by 11-20 minutes of post-exercise steam-room therapy. Participants are encouraged to exercise on their own (e.g., 1-2 days of aerobic and/or resistance training) but to refrain from unsupervised steam-room sessions or any other form of heat therapy.
  Other Names: STEAM
  Arms: Heat & Aerobic Training (HEAT) Condition
Behavioral: Exercise Only — Participants receive 42 supervised 50-minute, moderately intensive (50-75% max HR) aerobic exercise sessions (3 times per week), followed by 11-20 minutes of post-exercise sitting in the lobby of the fitness facility. Participants are encouraged to exercise on their own (e.g., 1-2 days of aerobic and/or resistance training) but to refrain from unsupervised steam-room sessions or any other form of heat therapy.
  Other Names: ExOnly
  Arms: Exercise Only

SUMMARY:
This study is intended for inactive, middle-aged adults with untreated pre-hypertension who live in the Urbana-Champaign area, who are interested in a comprehensive program designed to enhance physical activity & reduce blood pressure. All participants will be asked to engage in a program developed in accordance with American Heart Association's recommendations. Specifically, the program will encourage and support lifestyle behavior changes such as quitting smoking, eating heart-healthy food, and reducing excessive alcohol, in addition to weekly exercise. The exercise program will involve a 14-week aerobic training program (3 weekly sessions, scheduled at study participants' convenience), and 2 pre- and 2-post-testing sessions.

DETAILED DESCRIPTION:
Exercise has been associated with enhanced cognitive functioning. Several physiological mechanisms of change have been proposed, including increased blood-flow, vascular functioning, and neurological changes. Similar outcomes are also associated with partial-body and full-body heat therapy (e.g. steam-room or dry-sauna). The purpose of this study is to compare full-body HEAT treatments combined with exercise in a 14-week program to an exercise-only condition. The exercise program will involve moderate-intensity aerobic exercise training. All participants will also be asked to adhere to the American Heart Association's guidelines for reducing and controlling blood pressure, including increasing physical activity (at least 50 minutes, 3 times/week as part of our supervised training sessions), stopping smoking altogether, eating healthier (limiting sodium, eating fruit, veggies, low-fat dairy and lean protein, and reducing saturated fat and total fat), drinking less alcohol (1-2 drinks a day max) and achieving and maintaining a healthy bodyweight (striving for a body mass index between 18 and 25).

It is hypothesized that heat treatments combined with exercise will enhance the body's adaptive responses to exercise which in turn, should reduce blood pressure & blood flow, and improve cognitive functioning and related psychosocial outcomes (including anxiety and mindfulness). A two-armed (parallel groups design) randomized controlled trial involving heat and aerobic training (HEAT) will be compared with an exercise only (ExOnly) control condition. Therefore, the HEAT groups will receive 42 exercise classes each followed by a heat treatment involving 11-20 minutes of steam-room therapy. Post-exercise time will be matched in the control condition by having participants sit in the lobby after each session. The exercise interventions and assessments will be conducted by trained exercise staff. The participants will be assessed at baseline and post-intervention. Additionally, brief assessments will be administered at each session (pre and post) and logs will be administered to participants on a weekly basis. Assessments will include (a) physical activity & biometric monitoring, (b) performance on neurocognitive tests, (c) endothelial function, (d) a battery of psychosocial questionnaires, and (e) functional performance measures.

ELIGIBILITY:
Inclusion Criteria:

* Age 45 to 64
* Confirmed pre-hypertensive (120-139 mmHG Systolic / 80-89 Diastolic mmHG) blood pressure by our laboratory staff
* Low active (< 2 days per week for 30+ minutes over the past 3 months)
* Able and willing to try to adhere to American Heart Association guidelines for managing multiple lifestyle factors contributing to high blood pressure including increasing physical activity (at least 50 minutes, 3 times/week as part of our supervised training sessions), stopping smoking altogether, eating healthier (limiting sodium, eating fruit, veggies, low-fat dairy and lean protein, and reducing saturated fat and total fat), drinking less alcohol (1-2 drinks a day max) and achieving and maintaining a healthy bodyweight (striving or a body mass index between 18 and 25).
* Able to commit to the full length of our program without missing more than 2 consecutive weeks
* Capable of performing moderately intensive aerobic exercise
* Willing to be randomized to one of two groups
* Able to commute to and from fitness facility and UIUC campus
* Own smartphone and have reliable at-home internet access
* Have correctable vision (i.e., at least 20/40 with glasses or contacts with no color blindness)
* Not involved in regular weekly relaxation methods (e.g., yoga, meditation) or heat therapy (e.g., steam-room, sauna, hot baths)
* Not heat sensitive (e.g., have not experienced heat-induced severe rashes, pain, numbness, or tingling; experienced heat-related cramps, illness, or heatstroke; or had surgery requiring general anesthesia that has caused subsequent difficulty regulating body temperature)
* Do not have any type of neuropathy (e.g., peripheral, diabetic)
* Not depressed as indicated by a telephone screening (Abbreviated 5-item Geriatric Depression Scale; GDS-5 score < 2)
* No cognitive impairment as indicated by a telephone screening (Telephone Interview Cognitive Survey; TICS score > 21)

Exclusion Criteria:

* Too young (< 45) or too old (> 64)
* Normotensive (< 120 mmHG Systolic / < 80 Diastolic mmHG) or hypertensive (> 140 mmHG Systolic / > 90 Diastolic mmHG) blood pressure
* Too active (as defined by regularly exercise 2 or more days per week for 30+ minutes over the past 3 months)
* Unable or unwilling to comply with American Heart Association guidelines for managing multiple lifestyle factors contributing to high blood pressure including increasing physical activity (at least 50 minutes, 3 times/week as part of our supervised training sessions), stopping smoking altogether, eating healthier (limiting sodium, eating fruit, veggies, low-fat dairy and lean protein, and reducing saturated fat and total fat), drinking less alcohol (1-2 drinks a day max) and achieving and maintaining a healthy bodyweight (striving or a body mass index between 18 and 25).
* Unable to commit to full length of program
* Incapable of performing moderately intensive aerobic exercise
* Unwilling to be randomized to one of two groups
* Unable to commute to and from fitness facility and UIUC campus
* Does not own smartphone or have reliable at-home internet access
* Does not have correctable vision (i.e., at least 20/40 with glasses or contacts with no color blindness)
* Already involved in regular weekly relaxation methods (e.g., yoga, meditation) or heat therapy (e.g., steam-room, sauna, hot baths)
* Has heat sensitivity (e.g., heat-induced severe rashes, pain, numbness, or tingling; experienced heat-related cramps, illness, or heatstroke; or had surgery requiring general anesthesia that has caused subsequent difficulty regulating body temperature)
* Has any type of neuropathy (e.g., peripheral, diabetic)
* Has depression (as defined by GDS-5 score of 2 or higher)
* Has cognitive impairment (as defined by < 21 on TICS)

Ages: 45 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 41 (Actual)
Dates: Start 2015-08-21 (Actual); Primary Completion 2017-05-24 (Actual); Study Completion 2017-05-24 (Actual)

PRIMARY OUTCOMES:
blood flow | 14-week change
  Participants will be asked to fast for 6 hours and avoid alcohol & caffeine for 24 hours. They will arrive in a postprandial state and blood flow will be assessed on the calf using strain-gauge plethysmography. Data will be presented as peak hyperemic calf blood flow (CBF) and total CBF. Total CBF will be calculated as area under the curve of the 3-min hyperemic CBF response, based on 13 measures (post-occlusion) using the trapezoidal integration method (see Heffernan et al 2009). Total CBF is an overall estimate of the dilatory capacity of the vessels and therefore serves as an indirect measure of endothelial function.
blood pressure | 14-week change
  Resting systolic and diastolic will be assessed on the upper-arm with an automated Omron device that takes 3 continuous measurements and reports the average. After study enrollment, participants will be asked to avoid certain medications, foods and beverages known to alter these measurements. Upon entering the research site, participants will be instructed to sit quietly in a dimly lit room for 10 minutes prior to assessments. Staff will then assess blood pressure in three sequential positions (lying supine, sitting in chair, standing). The 14-week change in blood pressure will be defined as the difference between baseline and program end, using the average measures recorded at each position for systolic, diastolic, and mean arterial pressure.

SECONDARY OUTCOMES:
anxiety | 14-week change, intra-session change
  Perceptions of anxiety will be measured by the Hospital Anxiety and Depression Scale (HADS). Items for each subscale (anxiety and depression) will be summed (un-weighted) and averaged.
mindfulness | 14-week change
  The 15-item Mindfulness and Attention Scale (MAAS) will be used to assess mindfulness. A composite score will be computed based on an average of the unweighted sum of items.
stress | 14-week change, intra-session change
  Perceived stress will be assessed with the 10-item Perceived Stress Scale. A composite score will be calculated based on an unweighted sum and average of the items.
quality of life | 14-week change
  Quality of life will be measured by the 5-item Satisfaction with Life Scale. Items will be summed and averaged.
perceptions of memory | 14-week change
  Assessed by the 50-item Memory Self-Efficacy Questionnaire and the 12-item Memory Controllability Inventory. Items for each scale and subscale will be summed (un-weighted) and averaged. Scale composites will be used individually.
processing speed | 14-week change
  A linear combination (composite score based on an un-weighted sum) based on performance on the Digit Symbol Coding Task, Letter Comparison and Pattern Comparison will be used as an index of cognitive processing speed.
inhibition/attentional control | 14-week change
  A linear combination based on performance on standard Stroop and Flanker paradigms will be used as an index of inhibitory control. Established "cognitive cost" algorithms will be used incorporating only the difference in reaction times as one progresses to the most challenging trials. Scores will be weighed evenly across tests when calculating the composite index of inhibition/attentional control.
memory | 14-week change
  A linear combination based on performance on the N-back and Sternberg Task (working memory) as well as Logical Memory Test, Free Recall and Paired Associates (episodic memory) will be used as an overall index of memory ability. Reaction times will be weighed evenly across tests when calculating the composite measure. Only the most challenging trials of N-Back (2-back) will be used to compute an average reaction time score.
visual spatial skills | 14-week change
  A linear combination based on performance on the Card Rotations Test, Hidden Patterns Test, Spatial Relations, Paper Folding, and Form Boards will be used as an index of visio-spatial skills. Reaction times will be weighed evenly across tests when calculating the composite measure.
multi-tasking | 14-week change
  A linear combination based on performance on a Dual Task and Task-Switching paradigm will be used as an index of multi-tasking ability. The algorithm will use established measures involving cost in reaction times. Performance on both tests will be evenly weighted.
global executive functioning | 14-week change
  An iPad-version of the established Trail-Making (A&B) Test will be used to assess general executive functioning overall. The iPad version involves trials with stationary and moving stimuli within the A (alpha-only) and B (alpha-numeric) condition. A modified algorithm based on the commonly used index of global executive function (subtracting B - A) will be implemented for data analysis. Specifically, the outcome measure will be calculated as:
  Trails AB reaction time (RT) cost = ((Average RT for hard/moving B trials) - (Average RT for easy/stationary B trials)) - ((Average RT for hard/moving A - Average RT for easy/stationary A trials)).

CONTACTS AND LOCATIONS:
Overall Officials: Sean P Mullen, PhD, Principal Investigator — University of Illinois at Urbana-Champaign
Locations (1):
- Louise Freer Hall, Exercise Technology & Cognition Laboratory, Rm 253, Urbana, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Study Contact Form — http://exercisestudy.com/steam